CLINICAL TRIAL: NCT03796312
Title: The Effect of Tub Bathing and Sponge Bathing on Neonatal Comfort and Physiological Parameters in Late Preterm Infants: A Randomized Controlled Trial
Brief Title: The Effect of Tub vs Sponge Bathing on the Comfort of Premature Infants
Acronym: ComfortNEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tasdemir, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 455111
Record Dates: First submitted 2018-12-26; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Preterm Infant; Premature Birth
Keywords: Bathing; Comfort; Neonatal intensive care unit; Nursing care; Premature infant; Skin care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: A randomized controlled two-group pre-test and repeated post-test study design were adopted. Preterm infants were randomly allocated before bathing by the researcher using a random computer-generated table to one of two groups: sponge bathing (routine care) or tub bathing. The bathing procedures were performed by the researcher. Nurses and a second researcher were blinded to the study hypotheses.
Who Masked: Outcomes Assessor
Masking Description: Physiological data was collected by nurses trained by the lead researcher. Data on neonatal comfort behavior was collected by a second researcher and by research nurses who had been trained by the lead researcher. Those responsible for data collection were blinded as to the allocation of infants they were assessing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tub Bathing (Experimental): In this group, preterm infants were given tub bathing.
  Interventions: Behavioral: Tub Bathing
- Sponge Bathing (Active Comparator): Separate cotton cloths were prepared for each body area in the sponge bath. The room temperature was set to 26-27°C to prevent hypothermia. The temperature of the water used for sponge bathing was set to 37-38°C. Alongside the bath, the infant was placed on a flat, protected surface and washed from a bowl of water, using the same mild cleanser. The eyes, face, and head were wiped and dried while the baby was wrapped in a blanket. The wrap was opened so that body parts could be washed, dried, and then immediately rewrapped, after which infants were diapered.
  Interventions: Behavioral: Sponge Bathing

INTERVENTIONS:
Behavioral: Tub Bathing — The infant's face was washed and dried while still wrapped before being immersed. The water level in the tub was set at approximately 9-12 cm or deep enough to cover the baby's shoulders. A folded cloth towel was placed into the tub before bathing. The temperature of the bath water was controlled using a special water thermometer and adjusted to 37-38°C. The infant was held securely; the head and neck were supported on the researcher's forearm, and the shoulder was grasped using the researcher's thumb and finger. Cleaning was performed using a soft cloth and baby skin cleaner. The front and back areas were cleaned without turning the infant. The newborn was safely removed from the water and wrapped in a clean towel.
  Arms: Tub Bathing
Behavioral: Sponge Bathing — Sponge bathing is routine care of the clinic
  Arms: Sponge Bathing

SUMMARY:
The integumentary system protects the underlying body from the external environment, such as shocks, temperature, ultraviolet radiation, chemicals, and other threats. There is a considerable body of clinical evidence highlighting the importance of the stratum corneum and its barrier functions, which are especially beneficial for newborns. Given the dramatic transition from the aqueous womb to the dry terrestrial environment at birth, studies describing adaptations made by the skin barrier within the first month of life assume greater importance. The skin of the baby is morphologically and functionally different from the skin of adults. Neonatal skin is thinner, more fragile, and drier than adult skin; it is difficult to maintain fluid-electrolyte balance and temperature regulation. Notwithstanding, structure and function of skin continues to improve during the first months and even years of life. Special care procedures are nonetheless necessary to ensure healthy development, to protect the skin from irritation and reddening, and to help the newborn feel well. Therefore, this study, taking the form of a randomized controlled trial, aims to examine the effectiveness of tub bathing and sponge bathing on the physiological parameters (heart rate, respiration rate, oxygen saturation, body temperature) and comfort of late preterm infants. Increasing comfort and physiological stabilization in premature infants during neonatal care improves their neurophysiological development. Bathing procedures that support this development and will not expose the newborn to stress should be preferred.

DETAILED DESCRIPTION:
Increasing comfort and physiological stabilization in premature infants during neonatal care improves their neurophysiological development. Bathing procedures that support this improves and will not expose the newborn to stress should be preferred.This study aimed to examine the eﬀectiveness of tub bathing and sponge bathing methods on the comfort and physiological parameters of late preterm infants. The study was conducted in the Neonatal Intensive Care Unit of a university hospital in Turkey, between November 2015 and November 2016. Skin care is routinely performed between 08.00 and 09.00 in the form of sponge bathing. This research study sampled 120 stable, late preterm infants being cared for in the NICU. This sample was deemed adequate based on a sample size calculation conducted in PS Power and Sample Size Calculations (Version 3.0). Information concerning allocation was available only to the principal investigator. Participants were assigned a sequential number that was placed in an opaque, sealed envelope by the researcher who received the signed parental informed consent. When the participant was scheduled to be bathing, the envelope was opened by the researcher who then performed the test. The nurses could not be blinded to the allocation because of the nature of the intervention. However, the outcome assessment of the participants was blinded. Participats were randomly assigned to either sponge bathing or tub bathing groups. Bathing was performed anywhere from 6 to 48 hours post-birth, based on individual participant needs. Participants were subsequently placed in a preheated incubator, which varied according to the participant's weight and age. In order to compensate for such differences, the heads of all participants were placed at a height of 30 degrees in a right lateral position after bathing and they were monitored. The participants were not dressed during the observation period. After bathing, participants were left without intervention or contact for approximately 10 minutes or until settled before being assessed. The data collection instrument, the Preterm Infant Bathing Study Record, was designed specifically for this study. The instrument incorporates a number of scales for the measurement of outcome variables, physiological parameters, and demographic information (age, gender, type of delivery, gestational age, birth weight, body weight at study time, etc.). Outcome measures include neonatal comfort behavior and physiological parameters (body temperature, heart rate, oxygen saturation, respiratory rate). Those responsible for data collection were blinded as to the allocation of participants they were assessing. The ComfortNeo scale was used to measure newborns' comfort and pain intensity. Comfort was inferred based on infant behavior, which was evaluated on two separate occasions, 10 minutes before bathing and 10 minutes after bathing. Measurement took approximately 1-2 minutes. Internal consistency was measured by way of Cronbach's alpha coefficient, which was 0.94 before bathing, 0.93 after bathing for the second researcher, and 0.92 after bathing for the nurse. Kappa coefficients were approximately 0.84 for each sub-item. Thus, there was harmony between the two observers. Infant physiological parameters (heart rate, respiratory rate, oxygen saturation, and body temperature) were evaluated on three separate occasions (10 minutes before bathing, 15 minutes and 30 minutes after bathing).Statistical analysis was performed using SPSS 20.0 and SAS (ver.9.3), with statistical signiﬁcance set at p<0.05.

Data was presented as means and standard deviations for continuous variables, and frequencies for categorical variables. For participant characteristics, such as the type of delivery and sex, a Chi-square test was applied to determine whether there were signiﬁcant between-group differences. participant characteristics, such as birth weight and body weight at the time of the study, were evaluated for signiﬁcant between-group diﬀerences using a one way ANOVA test. For a comparison of the diﬀerent phases, measurement parameters (comfort score, heart rate, oxygen saturation, respiratory rate, body temperature) through the baths were averaged separately. Repeated measurement analysis of variance was performed to analyze both between and within-group diﬀerences, followed by the Bonferroni post-hoc test.

ELIGIBILITY:
Inclusion Criteria:

* All inborn infants with a gestational age of 34 weeks and 0 days to 36 weeks and 6 days (late preterm) were eligible to participate in this study.

Exclusion Criteria:

* Participants were excluded from the study if they were connected to
* a mechanical ventilator,
* if they had bathed in the last 12 hours,
* if within the first 78 hours of the postoperative period,
* had a central catheter,
* had received either a sedative and/or muscle relaxant,
* if they did not fulﬁll the inclusion criteria.

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Neonatal Comfort | An average of 1 year
  Data on comfort behavior was collected by a second researcher and by research nurses who had been trained by the lead researcher. Those responsible for data collection were blinded as to the allocation of infants they were assessing. The ComfortNeo scale was used to measure newborns' comfort. The ComfortNeo is a Likert-type scale consisting of six parameters: alertness, calmness/agitation, crying, body movement, facial tension, and (body) muscle tone. The lowest score that can be obtained using this scale is 6, and the highest score is 30. Scores in the range of 6 to 13 indicate that the newborn is comfortable, while scores 14-30 are indicative of pain or distress in the newborn, thus necessitating comforting. Comfort was inferred based on infant behavior 10 minutes before bathing and 10 minutes after bathing.

SECONDARY OUTCOMES:
Heart Rate | An average of 1 year
  The number of heartbeats per minute was obtained using a pulse oximetry device. A separate pulse oximetry probe was inserted into each of the infants.
Oxygen Saturation | An average of 1 year
  Oxygen saturation (SpO2) was obtained using a pulse oximetry device. A separate pulse oximetry probe was inserted into each of the infants. Pulse oximetry measures peripheral arterial oxygen saturation (%) as a surrogate marker for tissue oxygenation.
Respiration Rate | An average of 1 year
  The respiration rate is the number of breaths a person takes per minute. The rate is usually measured when a person is at rest and simply involves counting the number of breaths for one minute by counting how many times the chest rises.
Body Temperature | An average of 1 year
  Body temperature was measured using the axillary method (under the armpit)in degrees Celsius.

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz University Children's Health and the Nursing Department
Locations (1):
- Akdeniz Universty, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data sharing plans for the current study are unknown and will be made available at a later date

REFERENCES:
- [Background] Bryanton J, Walsh D, Barrett M, Gaudet D. Tub bathing versus traditional sponge bathing for the newborn. J Obstet Gynecol Neonatal Nurs. 2004 Nov-Dec;33(6):704-12. doi: 10.1177/0884217504270651. PMID 15561658
- [Background] Loring C, Gregory K, Gargan B, LeBlanc V, Lundgren D, Reilly J, Stobo K, Walker C, Zaya C. Tub bathing improves thermoregulation of the late preterm infant. J Obstet Gynecol Neonatal Nurs. 2012 Mar;41(2):171-179. doi: 10.1111/j.1552-6909.2011.01332.x. Epub 2012 Feb 29. PMID 22375955
- [Derived] Tasdemir HI, Efe E. The effect of tub bathing and sponge bathing on neonatal comfort and physiological parameters in late preterm infants: A randomized controlled trial. Int J Nurs Stud. 2019 Nov;99:103377. doi: 10.1016/j.ijnurstu.2019.06.008. Epub 2019 Jun 21. PMID 31442786